CLINICAL TRIAL: NCT06341478
Title: Understanding Tumor and Immune Dynamics and Predicting Response to Various Perioperative Therapies in Patients With Muscle-invasive Bladder Cancer
Brief Title: Investigator Grant (IG) 2022 27746
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Necchi, Professor, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IG-2022-27746
Record Dates: First submitted 2024-03-19; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Post-hoc biomarker analyses of ongoing phase 2 studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Radical cystectomy (Active Comparator): Radical cystectomy and pelvic lymphadenectomy upfront, according to the standar-of-care management
  Interventions: Drug: various neoadjuvant therapies
- Sacituzumab Govitecan (Experimental): SURE-01 trial: 4 courses of sacituzumab Govitecan, intravenously, at the dose of 7.5 mg/Kg on Day 1 and 8, every 21 days.
  Interventions: Drug: various neoadjuvant therapies
- Sacituzumab Govitecan + pembrolizumab (Experimental): SURE-02 trial: 4 courses of sacituzumab Govitecan, intravenously, at the dose of 7.5 mg/Kg on Day 1 and 8, every 21 days, added to pembrolizumab, intravenously, at the dose of 200 mg every 21 days, followed by radical cystectomy. After cystectomy, 13 courses of 200 mg pembrolizumab, intravenously, every 21 days.
  Interventions: Drug: various neoadjuvant therapies
- Nivolumab + abraxane (Experimental): NureCombo trial: 4 cycles of 360 mg nivolumab, every 3 weeks, added to nab-paclitaxel 125 mg/m2 on days 1 and 8, every 21 days, before radical cystectomy. After cystectomy, 13 courses of 360 mg nivolumab, intravenously, every 21 days.
  Interventions: Drug: various neoadjuvant therapies

INTERVENTIONS:
Drug: various neoadjuvant therapies — Radical cystectomy, Sacituzumab Govitecan (SG), SG + pembrolizumab, nivolumab+abraxane

SUMMARY:
Background:

Muscle-invasive bladder cancer (MIBC) is a systemic disease as >40% of patients (pts) ultimately develop recurrence after radical cystectomy (RC). For pts who cannot receive or refuse cisplatin-based chemotherapy there is no standard-of-care neoadjuvant therapy. Single-agent pembrolizumab, given neoadjuvantly in patients with T2-4N0M0 MIBC, documented a 42% pathologic complete response-rate (ypT0N0) in a previous AIRC-supported trial (PURE-01, NCT02736266; PMID: 30343614). However, there is a huge proportion of pts who do not benefit from single-agent immunotherapy. Antibody-drug conjugates (ADC) represent the next wave of MIBC treatment revolution. An umbrella of various neoadjuvant therapies including the ADC Sacituzumab govitecan (SG), SG plus pembrolizumab, and chemoimmunotherapy combination has been established to improve our knowledge on MIBC biology and to improve the outcomes.

Hypothesis:

By developing a robust biomarker program associated with therapeutic benefit of novel therapies or their combinations, along with an imaging biomarker development, the investigators will be able to identify suitable tumor characteristics for personalizing perioperative therapies in MIBC, coupled with the possibility to predict the pathological response to treatment.

Aims:

The project is aimed at characterizing the tumor and microenvironment characteristics of muscle-invasive bladder cancer, with a special focus on their changes induced by various neoadjuvant therapies preceding radical cystectomy.

The investigators will aim to evaluate the tumor and immune profile on matched pre- vs post-therapy samples and noninvasively monitor the response to treatment with the use of radiological assessments.

Experimental design:

The investigators will access tumor samples from matched pre-therapy (transurethral resection of the bladder tumor) and post-therapy (radical cystectomy) surgical interventions. They will also analyze the imaging analyses of combined bladder multiparametric MRI/Fluorodeoxyglucose Positron Emission Tomography (PET) scans pre-post neoadjuvant therapies, and will associate the data with the pathological response to treatment, expanding our previously reported work (PMID: 31882281).

Biomarker analyses will include the following: i.) multiplex immunofluorescence assays will allow the investigators defining the immune contexture of tumor lesion; ii.) multiparametric flow cytometry will allow the phenotypic and functional analysis of peripheral blood cells at single cell level; iii.) a whole transcriptome assay will enable investigators to assign specific molecular subtypes to pathological response and outcome, as previously reported (PMID: 33785257; 32165065).

Expected results:

The investigators will expect to identify the tumor characteristics and immune-profiling enabling them to delineate the selection of patients most suited for certain novel perioperative therapies, thus anticipating the developments in clinical research that are being conducted worldwide in MIBC.

The investigators will be also able to develop noninvasive tools for pathological complete response identification, thus enabling them to develop a next-generation of clinical trials aimed at sparing any radical local therapy on the bladder tumor.

Impact on cancer:

In principle, the present personalized strategy yields the potential to enhance the therapeutic standards achievable with RC alone as well as with single-agent immunotherapy and RC.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in NureCombo (NCT04876313), SURE-01 (NCT05226117), and SURE-02 (NCT05535218) clinical trials or candidates to radical cystectomy as per routine clinical practice.

  2. Histopathologically-confirmed urothelial carcinoma (UC). 3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1. 4. Clinical stage T2-T4N0M0, muscle-invasive bladder cancer (MIBC)

Exclusion Criteria:

1. Refusal to partecipate to the above studies
2. Unavailability of baseline tumor and blood samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Predictors of immune response to experimental combination therapies in MIBC. | Baseline (pre-therapy) to radical cystectomy
  Proportion of polymorphonuclear (PMN) cells, PMN-myeloid-derived suppressor cells (MDSCs), and intermediate monocytes (CD14+CD16+) in baseline blood samples of pathological complete responders compared to non-complete responders (pathological partial responders, pPR) and pathological nonresponders (pNR, ypT≥2N0 and ypN+).
Genomic predictors of response to experimental combination therapies in MIBC. | Baseline (pre-therapy) to radical cystectomy
  Proportion of gene mutations and fusions in baseline tumor samples of pathological complete responders compared to non-complete responders (pathological partial responders, pPR) and pathological nonresponders (pNR, ypT≥2N0 and ypN+).
Transcriptomic predictors of response to experimental combination therapies in MIBC. | Baseline (pre-therapy) to radical cystectomy
  Proportion of single gene or gene pathways signature scores in baseline tumor samples of pathological complete responders compared to non-complete responders (pathological partial responders, pPR) and pathological nonresponders (pNR, ypT≥2N0 and ypN+).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT06341478/Prot_000.pdf